CLINICAL TRIAL: NCT06784492
Title: Recovery After Acute Pulmonary Embolism
Brief Title: Incorporating Healthy Living Strategies to Aid in Recovery After Acute Pulmonary Embolism
Acronym: ERASE-PE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel Lachant, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009895; 1K23HL171867 (NIH)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Pulmonary Embolism
Keywords: Recovery acute pulmonary embolism; Six minute walk; Cardiac Effort; actigraphy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Living Intervention-1 (Experimental): Participants who receive daily messages about a healthy intervention.
  Interventions: Behavioral: Healthy Living Intervention-1
- Healthy Living Intervention-2 (Active Comparator): Participants who receive daily messages about a different healthy intervention.
  Interventions: Behavioral: Healthy Living Intervention-2

INTERVENTIONS:
Behavioral: Healthy Living Intervention-1 — Participants will receive a text or email each day with instructions about a healthy intervention.
  Arms: Healthy Living Intervention-1
Behavioral: Healthy Living Intervention-2 — Participants will receive a text or email each day with instructions about a healthy intervention.
  Arms: Healthy Living Intervention-2

SUMMARY:
The purpose of the ERAsE-PE study is to determine whether two different healthy living strategies (along with anticoagulation) might aid in recovery after a patient is hospitalized for pulmonary embolism. Specifically, Investigators will compare changes in Cardiac Effort (#heart beats used during the 6-minute walk test/walk distance) measured after an 8-week program.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking (>18 years old). Daily messages will be sent in English.
2. Acute PE with at least one of the following:

   1. any right ventricular enlargement or dysfunction on echocardiogram;
   2. CT Angiogram reporting any right ventricular enlargement; or
   3. elevated cardiac biomarker (NT-pro BNP or troponin above baseline). Criteria for enrollment will be included on source document.
3. Rate controlled atrial arrythmias (resting heart rate <110 beats/m) are eligible for enrollment. This includes atrial fibrillations. This is standard of care management for atrial fibrillation.
4. Subjects do need to take prescribed anticoagulation.

Exclusion Criteria:

1. Pregnancy.
2. Cardiac Effort >3.5 beats/m during 6MWT.
3. Resting tachycardia >110 beats/m at hospital discharge.
4. Chronic Thromboembolic Pulmonary Hypertension
5. Systolic blood pressure >180 mmHg at hospital discharge.
6. Inability to walk.
7. Estimated prognosis <12 months at the time of discharge due to underlying co-morbidities (e.g., cancer).
8. Advanced neurologic disease and would not be able to comply with the messages.
9. Lack of access to email or text messaging 10. Inability or unwillingness to follow daily instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in cardiac effort | Baseline and 3 months
  Change in cardiac effort is measured as the number of heart beats used during the 6-minute walk test.

SECONDARY OUTCOMES:
Mean number of health care visits (Health Care Utilization) | 3 months
  Subject medical records will be reviewed to determine the number of utilizations.
Mean change in Pulmonary Embolism Quality of Life Questionnaire (PEQOL) Score | baseline and 3 months
  The pulmonary embolism quality of life questionnaire ranges from 1 to 27, with higher scores indicating worse outcomes.
Mean change in 6 minute walk distance | baseline and 3 months
Mean change in activity as measured by Actigraph | baseline and 3 months
  The Actigraph triaxial accelerometer will be used to monitor the amount of activity taken at home on the non-dominant wrist. The accelerometer data will be downloaded and will include the amount of activity.
mean change in diagnoses | baseline and month 3
  Investifators will sum up the number of post-PE syndrome and CTEPH diagnoses and report the mean change in the sum between baseline and month 3.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes